CLINICAL TRIAL: NCT03304327
Title: Mindfulness and Yoga Training for Athletes With Concussion (MYTAC)
Acronym: (MYTAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: pro00086819
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Concussion
Keywords: Yoga; Mindfulness
MeSH Terms: conditions — Brain Concussion | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfullness and Yoga (Experimental): Subjects will receive yoga training either at their home or at the Center for Living Campus at Duke. Subjects will complete their yoga assignments for 5 consecutive days, along with a symptom checklist. On the 6th day, subjects will complete the symptom checklist and mail all checklists to the study team
  Interventions: Behavioral: Mindfulness and Yoga Training

INTERVENTIONS:
Behavioral: Mindfulness and Yoga Training — Centering and Breathing- Practice begins by turning attention to the breath to help participants make the transition from the busy, doing, outward focus of daily life into the mindful, balanced, internal focus central to yoga practice.
  Practices:Breath awareness, the relaxed abdominal breath. Posture Practice-Warm up with the range-of-motion sequence to take the major joints of the body through their full range of motion.This is done lying down with the head on the floor; the head can be supported by a small, folded towel if desired.
  Practices: Knee-to-chest sequence, Arms and Shoulders, Gentle Spinal Twist, Apanasana.
  Standing Poses for Strength and Balance, to enhance function and confidence. Practices: Mountain Pose, Flying Crane Sequence, Tree Pose, Warrior 2 and Side Angle.
  Relaxation- Practice concludes with guided relaxation to quiet the mind and calm the body.
  Practices: Seated Mountain Pose, even breath, extended exhalation,Yoga Nidra.

SUMMARY:
The purpose of this study is to establish the tolerability of mindfulness and yoga therapy in the post-concussion period.

DETAILED DESCRIPTION:
Athletes and patients aged 15 - 60 will receive standard sports concussion evaluations at the Duke Sports Science Institute (SSI) and will learn about the study by the primary clinicians evaluating sports concussion at the SSI. Subjects will receive yoga training either at their home or at the Center for Living Campus at Duke. Subjects will complete their yoga assignments for 5 consecutive days, along with a symptom checklist. On the 6th day, subjects will complete the symptom checklist and mail all checklists to the study team in a stamped envelope. We expect to enroll 20 subjects.

If a subject has significant worsening of their symptoms and wishes to discontinue the study, they are requested to contact the study PI, Joel Morgenlander, MD. At that time, Dr. Morgenlander will document the specific reasons for discontinuation of the protocol. All follow-up care for their concussion will be through the provider they are already seeing for concussion. There is no significant risk to the athlete for participation except possible transient increase in their concussion symptoms. Benefits include possible hastening of recovery from their concussive symptoms and receiving training in mindfulness and yoga from a certified yoga instructor.

ELIGIBILITY:
Inclusion Criteria:

* Injury sustained within 30 days of enrollment
* Being seen for concussion at the Sports Science Institute (SSI) at Duke University Medical Center
* living in a 30 mile radius of the SSI
* SCAT5 (Sport Concussion Assessment Tool 5) modified symptom checklist score of greater than 12

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Tolerability of mindfulness yoga therapy in the post-concussion period as measured by a rating scale. | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Joel Morgenlander, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No